CLINICAL TRIAL: NCT06396442
Title: Patient Worries Previous to Dental Treatment: a Multicenter Study
Brief Title: Patient Worries Previous to Dental Treatment
Status: Recruiting | Type: Observational
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, Principal Investigator, Aula Dental Avanzada
Other Study IDs: WORRIES
Record Dates: First submitted 2024-04-28; First posted 2024-05-02 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Patients
Keywords: dental treatment; worry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a multicenter cross-sectional study that aims to provide a snapshot of the experience of patients before starting dental treatment.

DETAILED DESCRIPTION:
Although the information is of limited duration, it could represent a descriptive view of a particular context of the dental profession in Spain. This qualitative information on patients' concerns may help the clinician to categorize patients' concerns, facilitate communication, and manage their expectations before initiating treatment.

Patients attending 6 different clinics in Spain consecutively for two years constitute the study sample. Questionnaires will be given to patients who consented to participate in the study, prior to the start of treatment. In addition to the questionnaire, additional demographic data will also be recorded.

The data will be analyzed statistically and appropriate conclusions will be drawn.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are going to receive dental treatment.

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who, after being informed about the treatment to be performed and about the research, agreed to answer the questionnaire would be included. The questionnaire should be answered just after receiving the clinical information on their treatment and before receiving the financial information on the treatment.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Worry or anxiety | Day 0
  Degree of concerns and anxiety the patient has prior to dental treatment by Numeric Rating Scale (NRS) form 0 to 10, being 0 "None" and 10 "Very much".
Fear of anesthesia | Day 0
  Degree of fear of anesthesia before undergoing dental treatment by Numeric Rating Scale (NRS) form 0 to 10, being 0 "None" and 10 "Very much".
Fear of pain | Day 0
  Degree of fear of pain before undergoing dental treatment by Numeric Rating Scale (NRS) form 0 to 10, being 0 "None" and 10 "Very much".
Fear of postoperative pain | Day 0
  Degree of fear of postoperative pain before undergoing dental treatment by Numeric Rating Scale (NRS) form 0 to 10, being 0 "None" and 10 "Very much".
Fear of chewing disability | Day 0
  Degree of fear of not being able to eat well after dental treatment by Numeric Rating Scale (NRS) form 0 to 10, being 0 "None" and 10 "Very much".
Treatment aesthetic effect | Day 0
  Degree of fear of the aesthetic effect that the treatment could have by Numeric Rating Scale (NRS) form 0 to 10, being 0 "None" and 10 "Very much".
Economic cost | Day 0
  Degree of fear of the economic cost of the treatment by Numeric Rating Scale (NRS) form 0 to 10, being 0 "None" and 10 "Very much".
Fear of contagion | Day 0
  Degree of fear of possible contagion during treatment by Numeric Rating Scale (NRS) form 0 to 10, being 0 "None" and 10 "Very much".

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Dental Esteve, Alicante, Alicante, Spain